CLINICAL TRIAL: NCT01872169
Title: Investigating the Prevalence of Disordered Eating in Children and Adolescents Attending the Great Ormond Street Gastroenterology Clinic
Brief Title: Investigating Prevalence of Disordered Eating in Children With GI Disorders
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was withdrawn prior to commencement
Sponsor: Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 13BS03
Record Dates: First submitted 2013-05-29; First posted 2013-06-07 (Estimated); Last update posted 2022-01-24 (Actual); Status verified 2013-06

CONDITIONS: Disordered Eating

ARMS (1):
- Disordered eating screening questionnaire (Other)
  Interventions: Other: Disordered eating screening questionnaire

INTERVENTIONS:
Other: Disordered eating screening questionnaire

SUMMARY:
Gastroenterological disorders are disorders affecting the stomach, intestines and associated organs. Symptoms of these types of disorders vary but often include vomiting, diarrhoea, weight loss and loss of appetite. Due to the nature and symptomatology of these disorders research has suggested that sufferers may be vulnerable to developing disordered eating behaviours. Treatment of such disorders often requires dietary restriction which has been found to lead to an obsessive preoccupation with food and in some cases to an increase in binge eating. Further to this, symptoms of Gastroenterological disorders such as vomiting have also been suggested to be linked with disordered eating. At the present there is limited research in this area and as such evidence is inconclusive. Particularly little research has looked at this area in relation to adolescents, who have been recognised as being at increased risk for the development of disordered eating . Gastroenterological disorders are likely to affect the typical development of eating habits and therefore it seems plausible they may also predispose adolescents to developing abnormal eating behaviours /weight concerns.

The aim of this study is to further investigate the possibility that Gastroenterological disorders may be a risk factor for disordered eating in children and adolescents. This study will recruit children/ adolescents aged 5-17 and their parents, who are attending Great Ormond Street Gastroenterology Clinic and ask them to complete a screening questionnaire. The recruitment process will be on going for around 5 months until the study has around 300 participants. Following this initial questionnaire, participants who are categorised as screening positively for disordered eating and a 10% sample of participants that screen negatively, will be contacted to complete a further questionnaire interview that will look more specifically into this area.

ELIGIBILITY:
Inclusion Criteria:

* Children/adolescents between the age of 5-17 and their parents who are attending the Gastroenterological Clinic. We will recruit all patients that fall within the age range, including both new patients and existing patients.

Exclusion Criteria:

* Parents/ adolescents unable to communicate English will be excluded from the current study.
* Children under the age of 5 and over the age of 17 will also be excluded.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2013-07 (Estimated); Primary Completion 2014-11 (Estimated); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
Disordered eating screening questionnaire | Questionnaire administered once after recruitment

SECONDARY OUTCOMES:
Developmental and Well Being Assessment | Administered once following inital screening

CONTACTS AND LOCATIONS:
Locations (1):
- Great Ormond Street Hospital, London, United Kingdom